CLINICAL TRIAL: NCT05763693
Title: Vitality in Infants Via Azithromycin for Neonates Trial
Acronym: VIVANT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21-34232
Record Dates: First submitted 2023-02-24; First posted 2023-03-10 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Neonatal Death; Infectious Disease; Nutritional Deficiency
Keywords: Low birth weight; underweight neonates
MeSH Terms: conditions — Perinatal Death; Communicable Diseases; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Azithro-Azithro (Active Comparator): A single oral dose of azithromycin (20 mg/kg) at baseline and a single oral dose of azithromycin (20 mg/kg) at the day 21 follow-up
  Interventions: Drug: Azithromycin at Baseline; Drug: Azithromycin at Day 21
- Azithro-Placebo (Active Comparator): A single oral dose of azithromycin (20 mg/kg) at baseline and a single oral dose of matching placebo at the day 21 follow-up
  Interventions: Drug: Azithromycin at Baseline; Other: Placebo at Day 21
- Placebo-Azithro (Active Comparator): A single oral dose of placebo at baseline and a single oral dose of azithromycin (20 mg/kg) at the day 21 follow-up
  Interventions: Drug: Azithromycin at Day 21; Other: Placebo at Baseline
- Placebo-Placebo (Placebo Comparator): A single oral dose of placebo at baseline and a single oral dose of matching placebo at the day 21 follow-up
  Interventions: Other: Placebo at Baseline; Other: Placebo at Day 21

INTERVENTIONS:
Drug: Azithromycin at Baseline — this group will be randomized to receive a single oral dose of azithromycin (20mg/kg) at baseline
  Arms: Azithro-Azithro; Azithro-Placebo
Drug: Azithromycin at Day 21 — this group will be randomized to receive a single oral dose of azithromycin (20mg/kg) at the day 21 visit
  Arms: Azithro-Azithro; Placebo-Azithro
Other: Placebo at Baseline — this group will be randomized to receive Placebo at baseline
  Arms: Placebo-Azithro; Placebo-Placebo
Other: Placebo at Day 21 — This group will be randomized to receive Placebo at the day 21 visit
  Arms: Azithro-Placebo; Placebo-Placebo

SUMMARY:
Nearly half of child deaths occur during the neonatal period, and 80% of those occur in babies with low birthweight. Although tremendous progress has been made towards reducing under-five mortality globally, declines in neonatal mortality lag behind those observed in older children. Low birthweight babies are at increased risk of poor outcomes compared to those who are term-appropriate for gestational age, including mortality, stunting, and growth failure. Recent evidence has demonstrated that the incidence of wasting and linear growth failure is highest between birth and 3 months of age, substantially earlier than previously thought. Interventions are urgently needed to improve outcomes in low birthweight babies; however, these interventions must not interfere with breastfeeding and thus some well-established interventions used to treat or prevent malnutrition in older children cannot be considered. The investigators recently demonstrated that biannual mass azithromycin distribution reduces all-cause childhood mortality by approximately 25% in infants aged 1-5 months, with stronger effects seen in underweight infants. This study did not include neonates due to the risk of infantile hypertrophic pyloric stenosis (IHPS) that has been hypothesized to be associated with macrolide use during early infancy. However, our study team documented only a single case of IHPS among 21,833 neonates enrolled in a trial of azithromycin versus placebo administered to neonates aged 8-27 days for prevention of infant mortality, documenting no major risk of IHPS associated with azithromycin. Here, the investigators propose an individually randomized trial where participants will receive a single oral dose of azithromycin (administered either during the neontal period or 21 days after enrollment), two does of oral azithromycin spaced 21 days apart, or two doses of placebo to evalute if azithromycin improves nutritional outcome and reduces infectious burden among neonates aged 1-27 days who are either low birthweight (<2500 g at birth) or underweight (weight-for-age Z-score < -2 at enrollment). The primary outcome will be weight-for-age Z-score at 6 months of age compared between arms. The investigators anticipate that the results of this study will provide definitive evidence on azithromycin as an early intervention for low birthweight/underweight neonates, who are at the highest risk of adverse outcomes.

DETAILED DESCRIPTION:
The Vitality in Infants Via Azithromycin for Neonates Trial (VIVANT) is a proposed 1:1:1:1 randomized placebo-controlled trial to determine whether a single oral dose of azithromycin (20 mg/kg) administered either in the early or late neonatal/early infancy period is effective for improving infant growth outcomes, and if there is additional benefit of administration of a second dose of azithromycin 21 days after the first dose (Figure 2). This intervention schedule will allow for several questions related to azithromycin administration in neonates to be answered efficiently, including:

1. A single oral azithromycin dose compared to placebo, administered either earlier or later during the neonatal period or early infancy.
2. Two oral doses of azithromycin spaced 21 days apart compared to placebo.
3. Two oral doses of azithromycin compared to a single oral dose of azithromycin, which would allow for determination of any dose-dependent effects.
4. An early dose of azithromycin compared to a later dose of azithromycin, which may be beneficial if administration of azithromycin earlier during the neonatal period increases risk of IHPS

ELIGIBILITY:
Inclusion Criteria:

* Aged 1-27 days old
* Birthweight < 2500 g and/or weight-for-height Z score <- 2 standard deviations at enrollment
* Weigh at least 1500 g at time of enrollment
* Able to feed orally
* Family intends to stay in the study area for at least 6 months
* Written informed consent from at least one caregiver
* Afebrile
* Caregiver at least 18 years old
* No known allergy to macrolides
* No hepatic failure manifested by neonatal jaundice
* Not currently an inpatient at the clinic
* Not being transferred to a hospital for clinical complications

Exclusion Criteria:

* Birthweight > 2500 g
* Weigh less than 1500 g at time of enrollment
* Unable to feed orally
* Family planning to move within 6 months
* Mother/ caregiver not willing to participate
* Allergic to macrolides
* Hepatic failure manifested by neonatal jaundice
* Currently being seen as an inpatient at the clinic
* Currently being transferred to a hospital for clinical complications

Ages: 1 Day to 27 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4000 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
weight gain at 6 month of age | 6 months
  Weight for Age Z score

SECONDARY OUTCOMES:
IHPS | 21 days
  Signs of IHPS will be screened at the 21 day follow up visit. diagnosed cases of IHPS will be reported by arm
Mortality at 6 months | 6 months
  Vital status will be verified at each follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Oldenburg, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- Centre de Recherche en santé de Nouna, Nouna, Burkina Faso

IPD SHARING:
Plan to Share IPD: No